CLINICAL TRIAL: NCT03714334
Title: Phase I Trial of DNX-2440 Oncolytic Adenovirus in Patients With Recurrent Glioblastoma
Brief Title: DNX-2440 Oncolytic Adenovirus for Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Break of stock
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: DNAtrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2440GBM1
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Glioblastoma; Glioblastoma, Adult
Keywords: Recurrent Glioblastoma; oncolytic virus; immunotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DNX-2440 injection (Experimental): all the patients included will be treated with the experimental agent
  Interventions: Drug: DNX-2440 injection

INTERVENTIONS:
Drug: DNX-2440 injection — DNX-2440 virus will be injected stereotactically

SUMMARY:
Patients with first or second recurrence of GBM will be treated with stereotactic injection of the oncolytic virus DNX-2440.

DETAILED DESCRIPTION:
After inclusion in the trial, stereotactic biopsy will be performed. In the same surgery, the experimental agent will be injected also by stereotactic system, in a different part of the lesion, in a region considered viable tumor, using a cannula especially designed for virus injection.

Follow-up will include clinical visits and MRI No other treatment for the tumor will be used until progression is documented. iRANO criteria and volumetric measurement of the tumor will be used.

Any further treatment after progression will be at the criteria of the treating physician

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to give informed consent.
2. Patient must be, in the investigator opinion, able to comply with all the protocol procedures.
3. Age ≥18
4. Negative pregnant test in case of fertile women*
5. Patients with diagnosis of first or second recurrence of Glioblastoma or any of its variants (Gliosarcoma, Giant cell Glioblastoma or epithelioid Glioblastoma) based on histopathology at first diagnosis and clinical and radiological follow-up. Recurrences within the radiation field will be considered if there is confirmed growing of the lesion in two MRI, or occur at least 12 weeks after completion of radiotherapy, or if there is clear histopathological confirmation of tumor recurrence. This limitation does not apply for recurrences occurring outside the radiation field
6. A single measurable lesion bigger than 10 mm in two perpendicular diameters, considered appropriate for safe stereotactic biopsy and virus injection without entering the ventricle.
7. No other chemotherapy or immunotherapy for the tumor in the four weeks previous to the inclusion
8. Karnofsky Performance Status ≥ 70 before inclusion.
9. Must have adequate renal, bone marrow and liver function.
10. Steroid-free or requiring stable doses of a maximum of 2mg dexamethasone /day or equivalent in the previous two weeks.

    * A woman is considered fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

1. Severe infections or intercurrent medical conditions including, but not limited to, severe renal, hepatic, heart or bone marrow failure, that, on investigator´s criteria, do not allow the inclusion. Patients must be afebrile at baseline [i.e., < 38 degrees (C)].
2. Patients with an enhancing lesion bigger than 25cc, including necrotic tumor portions encircled inside the enhancing areas.
3. Subjects with immunodeficiency, autoimmune conditions or active hepatitis.
4. Any medical or psychological condition that might interfere with the subject's ability to participate or give informed consent or would compromise the patient's ability to tolerate therapy or any disease that will obscure toxicity or dangerously alter drug metabolism.
5. Current diagnosis of other cancer except in situ cervical cancer, basal or squamous cell carcinoma of the skin. Patients with a history of another cancer remain eligible if they are cancer free for at least three years.
6. Pregnant or breast-feeding females will be excluded, due to the risk for the fetal development of a recombinant virus containing genes related to cellular growth and differentiation.
7. Severe bone marrow hypoplasia.
8. AST and/or ALT > 4 times over upper normal laboratory level
9. Neutrophils < 1.5 x 109/L
10. Thrombocytes ≤ 100 x 109/L
11. Hemoglobin < 9g/dl
12. Multiple lesions, extensive ill-defined diffuse lesions, or lesions considered risky for stereotactic injection of virus, like periventricular lesions.
13. Patients with Li-Fraumeni Syndrome or with a known germ line deficit in the retinoblastoma gene or its related pathways.
14. Biologic/immunotherapy (e.g., IL-2, IL-12, interferon) within 4 weeks of DNX-2440 administration.
15. Vaccination of any kind within 4 weeks prior to DNX-2440 administration.
16. Inability to undergo MRI examination for any reason.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events after brain administration of DNX-2440. | 8 weeks
  Incidence and severity of adverse effects will be collected and described

SECONDARY OUTCOMES:
Overall Survival at 12 months (OS12) | 12 months
  rate of patients surviving at 12 months since injection
Overall survival | 25 months
  Survival along the whole interval of follow-up
Overall response rate (ORR) | 6 months
  total of patients with Complete responses plus partial responses

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain